CLINICAL TRIAL: NCT02173795
Title: Berodual® Respimat® Inhaler Versus Berodual® MA Using HFA (Hydrofluoroalkane) 134a as Propellant in Adult Patients With Asthma, Chronic Obstructive Pulmonary Disease, or Mixed Conditions, an Open-label, Crossover Trial Over a 7-week Treatment Period With Each Formulation: ' A Study to Compare Patient Preference'
Brief Title: Berodual® Respimat® Versus Berodual® Metered Aerosol (MA) Inhaler in Patients With Asthma, Chronic Obstructive Pulmonary Disease, or Mixed Condition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 215.1357
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

ARMS (1):
- Berodual® Respimat® - Berodual® MA HFA (Experimental): randomized sequence
  1. Berodual® Respimat® (20 µg ipratropium bromide + 50 µg fenoterol hydrobromide per actuation for 49 days)
  2. Berodual® MA HFA (20 µg ipratropium bromide + 50 µg fenoterol hydrobromide per puff for 49 days)
  Interventions: Drug: Berodual® Respimat®; Drug: Berodual® MA HFA

INTERVENTIONS:
Drug: Berodual® Respimat®
Drug: Berodual® MA HFA

SUMMARY:
The primary objective of this study was to investigate patients acceptability / preference of Berodual® Respimat® inhaler as compared to the conventional Berodual® Metered Aerosol (MA) inhaler. Ease of handling and assembling the Respimat® inhaler at home under real life conditions was also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic obstructive pulmonary disease, asthma, or mixed conditions for a minimum of 6 months
* Male or female patients 18 years of age or older
* Patients who use at least 2 puffs t.i.d. of Berodual® MA HFA on regular use or at least 4 weeks prior to study
* Patients should be able to perform all study related tests including using a peak flow meter, to perform acceptable PEFR measurements, and should be able to maintain records (Patient Daily Diary Cards) during the study period as required in the protocol
* All patients must sign and Informed Consent Form prior to participation in the trial, i.e., prior to the run-in period in accordance with International Conference on Harmonisation (ICH) Good Clinical Practice (GCP)

Exclusion Criteria:

* Patients with significant disease other than chronic airways obstruction (CAO) will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Patients with a recent history (i.e., six months - or less) of myocardial infarction
* Patients with any cardiac arrhythmia requiring drug therapy or who have been hospitalized for heart failure within the past three years, including patients with hypertrophic cardiomyopathy and tachyarrhythmia
* Patients who regularly use oxygen therapy
* Patients with known active tuberculosis
* Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma are allowed
* Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis
* Patients who have undergone thoracotomy with pulmonary resection. Patients with history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1
* Patients with any upper or lower respiratory infection in the past six weeks prior to the screening visit (Visit 1) or during the run-in period
* Patients hospitalized or having had visits to the emergency room in the past six weeks before run-in period
* Patients who are currently in a pulmonary rehabilitation programme that will not be maintained throughout the duration of the study or who have completed a pulmonary rehabilitation programme in the six weeks prior to the screening visit (Visit 1)
* Patients with known hypersensitivity to anticholinergic drugs or any other components of the trial medication including excipients
* Patients medically treated for prostatic hyperplasia or bladder neck obstruction
* Patients with known narrow-angle glaucoma or raised intra-ocular pressure
* Patients who are being treated with beta-blocker medications Note: beta1-blocker eye medications for treatment of non-narrow angle glaucoma are allowed
* Patients using oral corticosteroid medication at unstable dose (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisolone per day or 20 mg every other day
* Patients on inhaled or short-acting beta-adrenergics other than the study medication
* Patients on inhaled or short-acting beta-anticholinergics other than the study medication
* Patients taking monoamine oxidase inhibitors
* Patients taking tricyclic antidepressants
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception for the previous three months (i.e., oral contraceptives, intrauterine inhalers, diaphragm or subdermal implants)
* Patients with a history of and/or active significant alcohol or drug abuse
* Patients who have taken an investigational drug within one month or six half-lives (whichever is greater) prior to the screening visit (Visit 1)
* Patients who have already been enrolled and randomised to a treatment group in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2002-10; Primary Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Patient's assessment of inhaler preference | Day 98
  patient preference questionnaire

SECONDARY OUTCOMES:
Rating of inhaler satisfaction | Day 49 and 98
  patient satisfaction questionnaire
Rating of willingness to continue using inhaler | Day 98
  patient preference questionnaire
Post-dose PEFRpm (Peak expiratory flow rate) | 30 minutes post-dose up to day 98
Retention of inhaler technique | day 49 and 98 (after 7 weeks of treatment)
  proficiency questionnaire
Use of rescue medication | up to day 98
Daytime and night-time symptom scores | up to day 98